CLINICAL TRIAL: NCT00185861
Title: Phase I Trial of Arsenic Trioxide and Stereotactic Radiotherapy for Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Cephalon (Industry); CTI BioPharma (Industry)
Responsible Party: Iris Catrice Gibbs, Principal Investigator, Stanford Univesity School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRNCNS0001; 79756; BRNCNS0001; NCT00185861
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Brain Cancer
MeSH Terms: conditions — Brain Neoplasms | interventions — Arsenic Trioxide; Radiosurgery

INTERVENTIONS:
Drug: Arsenic Trioxide
Procedure: Stereotactic radiosurgery

SUMMARY:
To investigate the safety of delivering arsenic trioxide (ATO) in combination with stereotactic radiotherapy in recurrent malignant glioma by performing an open label, Phase I dose escalation trial. Results from this study will provide a basis for further study of ATO combined with radiation therapy as a radiosensitizer for malignant brain tumors in future Phase II studies.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of recurrent disease.
* All patients will have received previous conventional radiotherapy at least 3 weeks prior to enrollment. Histologic verification of malignant glioma is required. If the initial primary brain tumor was histologically malignant glioma and subsequent contrast enhanced MRI imaging shows tumor consistent with recurrence, additional biopsy or surgery is not required. However, if a low-grade neoplasm was the initial histologic diagnosis, tissue confirmation of malignant glioma is required at the time of recurrence.
* Age: Patients must be >18 years of age
* Patients must have a Karnofsky >60%, and/or ECOG performance status <2
* Patients must have an estimated life expectancy of greater than 8 weeks.
* Patients must have normal organ and marrow functions as defined below:

  * Leukocytes >3,000/¼l
  * Absolute neutrophil count >1,500/¼l
  * Hemoglobin > 10 gm/dl
  * Platelets >100,000/¼l (transfusion independent)
  * Total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) <1.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits OR
  * Creatinine clearance >60mL/min/1.73 m2 for patients with creatinine levels above institutional normal
  * Serum potassium* e 4.0mEq/L
  * Serum magnesium* e 1.8mEq/L
  * Serum calcium* within the institutional normal range (should be corrected if low normal)
  * Electrocardiogram Normal
  * electrocardiogram with a rate corrected QT interval (QTc) <500 msec

    *Oral or intravenous supplementation may be used to normalize serum electrolytes
  * Phase I ATO Stereotactic Radiotherapy for Recurrent Malignant Glioma 16 of 44
* Informed consent All patients or their legal guardians must sign a document of informed consent indicating their understanding of the investigational nature of this study and the risks involved prior to any protocol related are performed (which does not include imaging and laboratory studies that help to establish eligibility).

Exclusion Criteria:- Patients who have had chemotherapy or conventional radiotherapy within 3 weeks of enrollment.

* Patients who have received prior radiosurgery or stereotactic radiotherapy within 10mm of the current target tumor.
* Patients may not be receiving any other investigational agents.
* Patients who cannot undergo MRI or CT are not eligible as MRI will be used to confirm the diagnosis and CT will be used for treatment planning.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to arsenic trioxide or other agents used in study.
* Patients who are taking substances known to prolong the QT interval, see Appendix B. If the QT prolonging drug is discontinued and switched to an alternative agent, the patients will be allowed to enroll into this protocol as long the agent has been discontinued for a period of at least 2 weeks.
* Patients currently taking Amphotericin B or related antifungal agents will be excluded due to potential for increased renal electrolyte wasting during arsenic trioxide therapy.
* Patients with known second-degree heart block or other cardiac dysfunction. New York Heart Association Class II or greater (see Appendix E)
* Uncontrolled intercurrent illnesses including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements. Phase I ATO Stereotactic Radiotherapy for Recurrent Malignant Glioma 17 of 44
* Patients must not be pregnant or breast-feeding. All patients with the potential for pregnancy should be counseled and requested to follow acceptable birth control methods (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Patients who are pregnant or breast-feeding will be excluded because no information on this agent exists with regard to safety of arsenic trioxide for a fetus or breast-feeding infant. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-12; Primary Completion 2008-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Describe and define toxicities of ATO combined with radiotherapy in patients with recurrent malignant glioma.
Define the maximum tolerated dose (MTD) of ATO combined with stereotactic radiotherapy for recurrent malignant glioma.

SECONDARY OUTCOMES:
Evaluate time to progression and survival
Evaluate radiographic tumor response rate
Determine the recommended dose for investigation in a Phase II study

CONTACTS AND LOCATIONS:
Overall Officials: Iris Catrice Gibbs, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States